CLINICAL TRIAL: NCT01921309
Title: Phase 3 Randomized Controlled Study to Demonstrate Safety and Effectiveness of the BIOLOX Delta CoC THR System
Brief Title: Trinity™ BIOLOX Delta™ CoC THR Multi-center Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: G120038; #G120038 (Other: IDE approved by CDRH)
Record Dates: First submitted 2013-06-10; First posted 2013-08-13 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; CDH
Keywords: osteoarthritis; avascular necrosis; rheumatoid arthritis; correction of functional deformity; dysplasia of the hip
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trinity CoC Total Hip System (Experimental): total hip replacement with a ceramic femoral head and ceramic acetabular cup liner
  Interventions: Device: Trinity CoC Total Hip System
- Trinity Ceramic-on-Poly THR (Active Comparator): total hip replacement with a ceramic femoral head and polyethylene acetabular cup liner
  Interventions: Device: Trinity Ceramic-on-Poly THR

INTERVENTIONS:
Device: Trinity CoC Total Hip System — total hip replacement with a ceramic femoral head which moves on a ceramic acetabular cup liner
  Arms: Trinity CoC Total Hip System
Device: Trinity Ceramic-on-Poly THR — total hip replacement with a ceramic femoral head which moves on a highly cross-linked ultra high molecular weight polyethylene acetabular cup liner
  Arms: Trinity Ceramic-on-Poly THR

SUMMARY:
To demonstrate the safety and effectiveness of the Trinity™ BIOLOX delta™ Ceramic-on-Ceramic Total Hip System in comparison to the Trinity™ Acetabular Hip System,which is FDA cleared for use in the U.S. The comparison will be based upon clinical success at the Month 24 endpoint.

DETAILED DESCRIPTION:
The clinical research results for the Trinity™ BIOLOX delta™ Ceramic-on-Ceramic Total Hip System will be compared to the control device

Clinical success is based upon Harris Hip Scores to evaluate functional status, adverse events, radiological assessments and no device failure (defined as removal, replacement, or modification of any device component).

ELIGIBILITY:
Inclusion Criteria:

1. preoperative Harris Hip Score of ≤ 70.
2. preoperative Harris Hip Total Pain score of at least moderate.
3. diagnosed with non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis, rheumatoid arthritis, correction of functional deformity, developmental hip dysplasia (DDH) and congenital hip dysplasia (CDH).
4. pain rating of none or slight and are at least 12 months post-operative in the contralateral hip, if applicable.
5. have sufficient femoral and acetabular bone stock as determined by a clinician, and are suitable to receive implants as confirmed by x-rays.

Exclusion Criteria:

1. have a nutritional problem (protein, calorie, or vitamin/mineral deficiency) that may impair wound healing mechanisms as determined by the clinician /investigator.
2. have a neurological disorders which may interfere or adversely affect gait, balance, or weight bearing (e.g. muscular dystrophy, multiple sclerosis).
3. diagnosed with metabolic disorders (e.g. osteomalacia), which may impair bone metabolism.
4. diagnosed systemic disease that would affect their welfare or the overall outcome of study (i.e. Paget's disease, renal osteodystrophy)
5. immunologically suppressed.
6. receiving systemic steroid therapy, excluding inhalers, within 3 months prior to surgery.
7. diagnosed Charcot's disease, metastatic or neoplastic disease.
8. evidence of active infections that may spread to other areas of the body (e.g. osteomyelitis, pyogenic infection of the hip joint, overt infection, untreated urinary tract infection, etc.).
9. presence of a previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) in the hip joint to be operated.
10. previous Girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.
11. diagnosed with systemic lupus erythematosus, pigmented villonodular synovitis, juvenile rheumatoid arthritis or other diagnoses with autoimmune etiology.
12. diagnosed with osteoporosis or as evidenced on a DEXA scan for males over 75 or females over 65 years of age (within the last 12 months).
13. require structural bone grafts in order to support the prosthetic component(s) or to shape the bone to receive the implant(s).
14. have acute femoral neck fracture or hip fractures.
15. have an above the knee amputation of the contralateral and/or ipsilateral leg.
16. have an existing total hip arthroplasty in the contralateral hip with a pain rating of 3 or more on a scale of 0 to 10, where 0 is "no pain" and 10 is "severe pain".
17. have had a total hip arthroplasty in the contralateral hip within the past 12 months.
18. have previously received a metal-on-metal hip arthroplasty.
19. have a highly communicable disease or diseases that may limit follow-up (e.g. immunocompromised conditions, hepatitis, active tuberculosis, etc.).
20. have any known sensitivity to device material.
21. Females who are pregnant.
22. Patients who are prisoners.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2012-12; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Success | 24 months post-operative
  * HHS ≥ 80 at Month 24 (good/excellent)
  * No serious, definitely device related complications with onset on or prior to Month 24
  * No radiographic failure at Month 24
  * No removal, replacement, or modification of any component on or prior to Month 24.

SECONDARY OUTCOMES:
HHS | 24 months post-operative
  • Individual components of the Harris Hip Score (total score, pain and function).
HOOS score | 24 months
  Hip injury and Osteoarthritis Outcome Score (HOOS).
Subjective pain | 24 months
  VAS pain score
survival | 24 months
  Kaplan-Meier survival curve
adverse events | 24 months
  Summary of device-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Trier, Ph.D., Study Director — Corin
Locations (10):
- United States (9):
  - Arkansas Specialty Orthopaedics, Little Rock, Arkansas
  - Denver Hip and Knee, Inc., Parker, Colorado
  - Connecticut Joint Replacement Institute (CJRI), Hartford, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Orthopaedic Institute, Tampa, Florida
  - FMC Orthopedic Division, Tampa, Florida
  - Resurgens Orthopaedics, Austell, Georgia
  - OrthoCarolina Hip & Knee Center, Charlotte, North Carolina
  - Memorial Bone & Joint, Houston, Texas
- Elective Orthopaedic Centre, Epsom, Surrey, United Kingdom